CLINICAL TRIAL: NCT03561428
Title: Discovery and Validation of Biomarkers of Lichen Sclerosus
Brief Title: Biomarkers of Lichen Sclerosus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Center for Vulvovaginal Disorders (Other)
Collaborators: Gynecologic Cancer Research Foundation (Other); George Washington University (Other)
Responsible Party: Principal Investigator, Andrew T. Goldstein, MD, Study Investigator, Center for Vulvovaginal Disorders
Other Study IDs: 091739
Record Dates: First submitted 2018-01-02; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Lichen Sclerosus
Keywords: lichen sclerosus
MeSH Terms: conditions — Lichen Sclerosus et Atrophicus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — All samples obtained in this study will be processed for RNA, protein and DNA extraction, which will be used for gene expression analysis. The samples collected will be snap-frozen in liquid nitrogen before transporting, and store in a -80C degree freezer in the Department of Medicine at the George Washington University School of Medicine in Ross Hall for a period of 5 years for further verification studies if needed, and then they will be destroyed unless the patient has consented to future research on their samples. The patient's name will not be on these specimens, but will instead be given a study number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lichen sclerosus (LS) is a skin condition of the external genitals (vulva) of women. LS causes vulvar itching, pain, and burning. In addition, LS causes scarring of the vulva which may cause significant lack of sexual pleasure or pain. Lastly, 4-6% of women with LS will develop vulvar cancer. The purpose of this study is to learn the gene expression file changes in skins affected by LS as compared to normal skins in order to discover the mechanism of the LS, and further to develop effective drugs to treat the condition.

DETAILED DESCRIPTION:
Lichen sclerosus (LS) is a chronic, lymphocyte mediated cutaneous disorder affecting approximately one in seventy women. Presenting symptoms may include intense pruritis, pain, burning, and dyspareunia. This disorder may affect any area of the skin, but has a notable predilection for the female genital region, in particular, the vulva, per anal area and the groin. Affected females outnumber affected males by 13:1. Typically, the patient is a menopausal woman, but prepubertal girls and women of all ages may be affected. The typical lesions of lichen sclerosus are white plaques and papules, often with areas of ecchymosis, excoriation, and ulceration. Often, there is destruction of the vulvar architecture with scarring of the clitoral prepuce, resorption of the labia minora, and narrowing of the introitus. Vulvar lichen sclerosus has a 4%-6% transformation malignant rate and women with the disease are at a 250-fold increased risk for developing vulvar carcinoma than women without lichen sclerosus. While the exact etiology of LS is as yet unknown, there is at least a suggested genetic component as evidenced by case reports of familial LS, findings of associations with HLA antigens, and high rates of concordance with other autoimmune disorder.

The purpose of this study is to determine the differences in the genomic/proteomic profiles between LS and normal skin biopsies for women with active vulvar lichen sclerosus in order to identify potential biomarkers that can be used for the prevention, early diagnosis and effective treatment for LS. The study will aim to identify genes/proteins/glycoproteins biomarkers that are associated with LS, select biomarkers associated with LS either individual candidate biomarker or as a panel, validate the identified candidate biomarkers for LS using targeted analysis of candidate biomarkers from independent LS specimen sets, develop assays to determine the clinical utilities of the identified biomarkers as minimum invasive tests for the early detection of LS and determine the clinical utility of biomarkers for biopsy-based tissue tests for LS diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 of age
* Diagnosis of active, Histologically proven, vulvar lichen sclerosus

Exclusion Criteria:

* Under the age of 18 or over the age of 75.
* Participants who are pregnant at the time of recruitment
* If, in the clinical opinion of Dr. Andrew Goldstein, she:

  * does not have active LS
  * has active infection
  * has evidence of any other dermatologic disease of the vulva
  * has evidence of neoplastic disease of the vulva
* If, in the opinion of Dr. Andrew Goldstein, they will be unable to keep the biopsy sites clean until they heal.
* If the biopsy specimen sent to dermatopathology is not confirmatory for active lichen sclerosus then the specimens obtained from that patient will be excluded from the study.

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The total number of subjects to expected to be recruited are 58 total.
  * six families with 2-3 family members affected in each family with LS
  * 40 patients (sporadic) with active lichen sclerosus
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-11-26 (Estimated); Study Completion 2019-11-26 (Estimated)

PRIMARY OUTCOMES:
Differential gene expression between LS and normal vulvar skin tissue | 1-2 year
  Gene expression obtained from biopsies via Next Generation Sequencing (RNASeq)
Differential protein expression between LS and normal vulvar skin tissue | 1-2 year
  Protein expression obtained from biopsies via Western blot
Identification of tissue-derived glycoproteins in serum | 1-2 years
  Glycoproteins identified via glycoproteomic technologies

CONTACTS AND LOCATIONS:
Overall Officials: Charles Macri, MD, Principal Investigator — George Washington University School of Medicine and Health Sciences; Sidney Fu, MD, PhD, Principal Investigator — George Washington University School of Medicine and Health Sciences; Andrew T Goldstein, MD, Principal Investigator — The Center for Vulvovaginal Disorders
Locations (1):
- The Centers for Vulvovaginal Disorders, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
The data will be summarized in publication and presentation. Individual results will not be communicated, and nor the study participants will be contacted about their results.

REFERENCES:
- See also: Informed Consent — http://cvvd.org/research